CLINICAL TRIAL: NCT02500290
Title: Antiplatelet Therapy in Acute Coronary Syndrome (ACS). Safety and Efficacy of Switching Antiplatelet
Brief Title: Antiplatelet Therapy in Acute Coronary Syndrome(ACS). Safety and Efficacy of Switching Antiplatelet
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fundación Pública Andaluza Progreso y Salud (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Other Study IDs: FPS-AAS-2014-01
Record Dates: First submitted 2015-07-07; First posted 2015-07-16 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-02

CONDITIONS: Acute Coronary Syndrome
Keywords: ACS
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute coronary syndrome

SUMMARY:
This study aims to describe antiplatelet therapy in ACS in Andalusia and make an assessment of efficacy and safety of hospital use Prasugrel / ticagrelor vs. Clopidogrel and Prasugrel switching to / ticagrelor patients pretreated with clopidogrel.

DETAILED DESCRIPTION:
The management of acute coronary syndrome has changed in recent years as reflected in the new Clinical Practice Guidelines of the European Society of Cardiology for the management of ACS with or without ST segment elevation, with the development and increased accessibility of the angiography and percutaneous coronary intervention and the arrival of the new antiplatelet (Prasugrel and Ticagrelor).

The ACS encompasses several clinical entities where dual antiplatelet therapy remains the basis of antiplatelet therapy and one of the mainstays of treatment. But the emergence of Prasugrel and Ticagrelor have changed the classical management with aspirin plus clopidogre

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the Coronary Care Unit at the time defined with an initial diagnosis of ACS.

Exclusion Criteria:

* Myocarditis, Takotsubo syndrome, pulmonary thromboembolism.
* Secondary MI or type 2, caused by an increase in demand or decrease oxygen (anemia, tachycardia, hypotension, heart failure, etc.). 11
* Patients under 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with acute coronary syndrome
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2014-11; Primary Completion 2019-02-21 (Actual); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
type of antiplatelet were used | 12 months
  There are the following therapeutic groups:
  Clopidogrel; Prasugrel; Ticagrelor; Switching to Prasugrel ; Switching toTicagrelor

SECONDARY OUTCOMES:
ischemic events after ACS during hospitalization | 3, 6 and 12 months
  Ischemic event is defined as the combined end point of stroke, reinfarction, stent thrombosis, restenosis and stent injury retreat previously treated
  1. thrombotic complications: stroke, stent restenosis, retreat of the culprit vessel, stent thrombosis, CVA
Total rate of hemorrhage and severity thereof under TIMI9 and BARC15 classification. Also it included as a safety endpoint all-cause mortality. | 3, 6 and 12 months
  bleeding complications: BARC, TIMI classification, transfusions, major bleedingbleeding complications: BARC, TIMI classification, transfusions, major bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Almedro Delia, MD, Study Director — Hospital Universitario Virgen Macarena
Locations (8):
- Spain (8):
  - Hospital de Jerez, Cadiz
  - Hospital de Puerto Real, Cadiz
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital de Antequera, Málaga
  - Hospital Regional de Málaga, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen Macarena, Seville

REFERENCES:
- [Derived] Almendro-Delia M, Padilla-Rodriguez G, Hernandez-Meneses B, Blanco-Ponce E, Arboleda-Sanchez JA, Rodriguez-Yanez JC, Soto-Blanco JM, Fernandez-Garcia I, Castillo-Caballero JM, Garcia-Rubira JC, Hidalgo-Urbano R. Nonadherence to ticagrelor versus clopidogrel and clinical outcomes in patients with ACS. Results from the CREA-ARIAM registry. Rev Esp Cardiol (Engl Ed). 2024 Feb;77(2):113-124. doi: 10.1016/j.rec.2023.05.011. Epub 2023 Sep 29. English, Spanish. PMID 37573968
- [Derived] Almendro-Delia M, Blanco-Ponce E, Carmona-Carmona J, Arboleda Sanchez JA, Rodriguez Yanez JC, Soto Blanco JM, Fernandez Garcia I, Castillo Caballero JM, Garcia-Rubira JC, Hidalgo-Urbano RJ. Comparative Safety and Effectiveness of Ticagrelor versus Clopidogrel in Patients With Acute Coronary Syndrome: An On-Treatment Analysis From a Multicenter Registry. Front Cardiovasc Med. 2022 May 27;9:887748. doi: 10.3389/fcvm.2022.887748. eCollection 2022. PMID 35711382